CLINICAL TRIAL: NCT02361853
Title: The Role of Immature Myeloid Cells, Monocytes, Dentritic Cells and Neutrophils in Human Pregnancies as Markers for Mature Pregnancy and Spontaneous Labor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0086-14-HYMC
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Parturition
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Active labor at term: Women in active labor normal pregnancy at term
  Interventions: Other: Exposure: abundance of Immature Myeloid Cells counts in blood samples; Other: Exposure: abundance of Immature Dentritic Cells counts in blood samples; Other: Exposure: abundance of Immature monocytes counts in blood samples; Other: Exposure: abundance of Immature neutrophils counts in blood samples
- Non-active labor at term: Women, normal pregnancy at term who come for usual follow up without signs for labor ( contraction / "show" discharge/ rupture of membranes).
  Interventions: Other: Exposure: abundance of Immature Myeloid Cells counts in blood samples; Other: Exposure: abundance of Immature Dentritic Cells counts in blood samples; Other: Exposure: abundance of Immature monocytes counts in blood samples; Other: Exposure: abundance of Immature neutrophils counts in blood samples
- Active labor, pre-term: Women in active pre term labor (34- 37w) normal pregnancy.
  Interventions: Other: Exposure: abundance of Immature Myeloid Cells counts in blood samples; Other: Exposure: abundance of Immature Dentritic Cells counts in blood samples; Other: Exposure: abundance of Immature monocytes counts in blood samples; Other: Exposure: abundance of Immature neutrophils counts in blood samples

INTERVENTIONS:
Other: Exposure: abundance of Immature Myeloid Cells counts in blood samples
Other: Exposure: abundance of Immature Dentritic Cells counts in blood samples
Other: Exposure: abundance of Immature monocytes counts in blood samples
Other: Exposure: abundance of Immature neutrophils counts in blood samples

SUMMARY:
Accumulating evidence suggest that the proliferative, invasive, and immune tolerance mechanisms that malignant tumors use to establish a nutrient supply and evade or edit the host immune response are similar to those used by the developing placenta during normal pregnancy. In addition to the shared capacity for invading through normal tissues, both cancer cells and cells of the developing placenta create a microenvironment supportive of both immunologic privilege and angiogenesis.

CD11b+Gr1+ cells are a heterogeneous population of bone marrow-derived cells (BMDC) that consist of immature myeloid cells (IMCs), and were first described as myeloid-derived suppressor cells. In healthy individuals, IMCs that are generated in the bone marrow differentiate into mature granulocytes, macrophages, or dendritic cells (DCs). These cells have been shown to play an essential role in mediating immune suppression in animal models of human tumors. As a result of tumor-induced alterations in myelopoiesis, IMCs have been found in peripheral blood, lymphoid organs and the tumor tissue itself. An increased population of IMCs was identified in patients with several tumor types. Accordingly, IMCs detected in the peripheral blood of such patients bearing express the common myeloid marker CD33 but lack markers of mature myeloid cells such as the MHC class II molecule HLADR.

IMCs have been shown to actively promote tumor growth and metastasis by modulating the cytokine environment, and through vascular remodeling by promoting angiogenesis.

It has been demonstrated in our laboratory that IMCs infiltrate placentas of pregnant mice and actively promote angiogenesis. These cells show striking similarity to IMCs that populate malignant tumors. Accordingly, human placentas are also infiltrated by a significant population of IMCs. Immunostaining of human placentas showed that IMCs comprise around 25% ( range 10-40%) of total placental CD45+ bone marrow-derived hematopoietic cells and that this population is located close to blood capillaries. The investigators also demonstrated that immature DCs, cells originally described to regulate the adaptive immune response, also promote angiogenesis in models of choroidal neovascularization, endometriosis and tumors.

Tho objective in this proposed study is to compare the abundance of IMC, DC, monocytes and neutrophils counts in blood samples of normal pregnancies: 1. in women in term active labor. 2. In women not in labor. 3. In pre term labor.

According to our previous findings, the investigators hypothesize that IMC's, monocytes and in active delivery (both term and pre term) will be lower than women without signs for labor. The investigators also hypothesize that DC's and neutrophils will be more abundant in active delivery (in term and pre term) than women without signs for labor.

Experimental plan:

Blood count will be collected from pregnant women who agree to participate in the research:

The samples will be sent for the routine complete blood count in Hillel Yaffe hematologic lab and also will be analyzed for IMC's and DC's population in our lab using fluorescent immunostaining with specific monoclonal antibodies and flow cytometry.

IMC's per total CD45 positive hematopoietic cells from the placental tissue will be analyzed using fluorescent immunostaining with specific monoclonal antibodies and flow cytometry . The specific location of these cells in the placenta will be identified within the placental tissue using Immunohistochemistry (IHC). The expression of pro angiogenic genes will be analyzed by RT PCR and Western blotting.

ELIGIBILITY:
Inclusion Criteria:

* Women in active labor normal pregnancy at term.
* Women, normal pregnancy at term who come for usual follow up without signs for labor ( contraction / "show" discharge/ rupture of membranes).
* Women in active pre term labor (34- 37w) normal pregnancy.

Exclusion Criteria:

* Unwilling of the women to participate in the research
* Signs for infection ( fever >38)
* Women in pre-term birth under 34 weeks.
* Administration of Celeston in 2 weeks prior to enrollment.
* Any complication to the women or fetus which require induction of labor ( Pre-eclampsia, Gestational Diabetes Mellitus A2, pre gestational diabetes, Intrauterine Growth Restriction).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women from: 34 weeks to 42 weeks
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Spontaneous labor | maximum two weeks